CLINICAL TRIAL: NCT05515965
Title: Acute Effect of Kinesiotaping Applied to the Thumb in Patients With Rheumatoid Hand
Brief Title: Kinesiotaping Applied to the Thumb in Rheumatoid Hand
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Arel University (Other)
Responsible Party: Principal Investigator, Ozge Baykan Copuroglu, Prelector/ Physiotherapist, Istanbul Arel University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RomatolojiParmak
Record Dates: First submitted 2022-08-24; First posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-08

CONDITIONS: Rheumatoid Arthritis; Kinesiotape; Hand Deformity
Keywords: Rheumatoid Arthritis; Kinesiotape; Grip Strength; Hand function; Hand deformity
MeSH Terms: conditions — Arthritis, Rheumatoid; Hand Deformities | interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinding was ensured by patients and rheumatologist were unaware the type of physiotherapy treatment application
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotape (Experimental): The patients in the Kinesiotape group were taped with the mechanical correction method.
  Interventions: Other: Kinesiotaping
- Control (Sham Comparator): In the patients in the Control group were taped with tensionless gluing of the I tape.
  Interventions: Other: Sham

INTERVENTIONS:
Other: Kinesiotaping — The mechanical correction method of taping to the Kinesiotape group was used. In rheumatoid hand patients, due to the presence of a deformity called hitchhiker's finger, the thumb is taped with 50-75% tension to create a pulling force in the direction of flexion and abduction. The application was performed with the patient in a sitting position with his arm supported by a pillow from the elbow. Evaluation parameters were evaluated before and 1 hour after the application, and the acute effect was examined. Both the dominant and nondominant hands of the patients were taped and the differences between the two hands were also examined.
  Arms: Kinesiotape
Other: Sham — Sham application was applied to both dominant and nondominant hands in Control Group patients. Sham taping is the bonding of I tape to the 1st finger without tension and does not contain any features. Evaluation parameters were evaluated before and 1 hour after the application, and the acute effect was examined. Both the dominant and nondominant hands of the patients were taped and the differences between the two hands were also examined.
  Arms: Control

SUMMARY:
Objective: It was aimed to evaluate the acute effect of Kinesiotape taping on pain, function, range of motion and grip strength parameters in patients with rheumatoid arthritis and hand involvement.

Material and Methods: A total of 34 patients, 27 women and 7 men, diagnosed with RA according to the American Rheumatism Association (ACR) criteria were included in our study. All patients were divided into two groups as Kinesiotape and Control groups, each consisting of 17 patients. Subjective pain intensity was evaluated with the Visual Analog Scale, range of motion was evaluated with a goniometer, functional evaluation was evaluated with the Grip Skill Test, hand grip strength was evaluated with a dynamometer, and finger grip strength was evaluated with a pinchmeter. Evaluation parameters were evaluated before and 1 hour after the application, and the acute effect was examined. The patients in the kinesiotape group were taped with the mechanical correction method and the patients in the Control group were taped with tensionless gluing of the I tape. Applications were made on both dominant and nondominant hands.

DETAILED DESCRIPTION:
This study is a double-blind, randomized clinical trial conducted by the Non-Interventional Ethics Committee from April 2018 to October 2018 in the Rheumatology unit of a university hospital in Turkey. The patients were divided in two groups using simple randomization method. There are 17 patients in groups. As the evaluation content; Socio-demographic information was recorded. Pain assessment was done by participants' subjective pain intensity Visual Analogue scale, mobility assessment was made by evaluating the range of motion with a goniometer, functional assessment was by grasping skill test, hand grip strength was measured by dynamometer, and finger grip strength was measured by pinchmeter. In our study, the mechanical correction method of taping to the Kinesiotape group was used. In rheumatoid hand patients, due to the presence of a deformity called hitchhiker's finger, the thumb is taped with 50-75% tension to create a pulling force in the direction of flexion and abduction. Sham application was applied to both dominant and nondominant hands in Control Group patients. Sham taping is the bonding of I tape to the 1st finger without tension and does not contain any features. Both the dominant and nondominant hands of the patients were taped and the differences between the two hands were also examined.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed as Level 2-3 Rheumatoid Arthritis
* no change in pharmacological treatment until 1 month before the study

Exclusion Criteria:

* Presence of acute disease
* Diagnosis of Level 4 Rheumatoid Arthritis
* Intra-articular or intramuscular injection application in the previous months
* Presence of hand-wrist surgery history in the last 6 months
* Non-rheumatoid hand deformity

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 34 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-10-01 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Subjective Pain Intensity | 1 hour
  The subjective pain intensity of the patients was assessed with the Visual Analogue Scale. The Visual Analog Scale includes scoring between 0 and 10. The corresponding numbers from 0 to 10 were explained to the patients. It was explained that the absence of pain was 0, the most severe pain felt was 10, and moderate pain was 5.
Range of Motion | 1 hour
  The range of motion of hand and metacarpophalangeal jonit were assessed using a goniometer
Functional Assessment | 1 hour
  Grip Skill test will also be applied, and this test was basically developed for cases with RA. It has three main components; Filling the glass with water, holding socks, envelopes with paper clips. The maximum time allocated to each test is 60 seconds. The time to complete the first and second tests is multiplied by 1.8 and added to the other values. The total score range is 10-279. A high score means impaired hand function. The mean score value in healthy individuals is 16.5 (11-20).
Hand muscle strength | 1 hour
  Hand grip strength was measured by dynamometer. The patient squeezed and released the dynamometer 3 times and the average of these three values was recorded.
Finger muscle strength | 1 hour
  Finger grip strength was measured by pinchmeter. The patient squeezed and released the dynamometer 3 times and the average of these three values was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Ozge Baykan Copuroglu, MSc, Principal Investigator — Istanbul Arel University
Locations (1):
- Ozge Baykan Copuroglu, Bahçelievler, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided